CLINICAL TRIAL: NCT05559034
Title: Identification of a Brain Oxygenation Marker for Cognition Using Functional Near Infrared Spectroscopy in Healthy Adults
Brief Title: Brain Oxygenation Marker for Cognitive Function in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor
Other Study IDs: 2205NR
Record Dates: First submitted 2022-09-12; First posted 2022-09-29 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Mental Fatigue
Keywords: Cortical tissue oxygenation; Cognition; Time-on-task; Functional Near Infrared Spectroscopy
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: The study will comprise only one group of healthy adults subject to a same behavioral and cognitive intervention.
  Interventions: Behavioral: Cognitive intervention

INTERVENTIONS:
Behavioral: Cognitive intervention — This is a cognitive intervention consisting in the repetition according to three blocks, of cognitive tasks (Stroop and N-back tasks) at variating workload levels (low, middle and high levels). Each cognitive task will be presented for each workload level during three minutes.

SUMMARY:
This study aims to identify a cortical oxygenation marker for cognitive function using functional Near Infrared Spectroscopy in healthy adults.

DETAILED DESCRIPTION:
This study will aim to establish a model between the cortical oxygenation and cognitive performances given modulations by experimental conditions including the cognitive workload and the time-on-task, and individual variabilities such as the age or the gender.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females 25-45 years old
2. BMI between 18.5 kg/m2 and 29.9 kg/m2
3. Conditions for study procedure compliance:

   * Willing and able to sign an informed consent form
   * Be fluent in English (self-reported C1 or C2 English level)
   * Be able to provide a cortical oxygenation signal (based on feasibility to fix the measurement device on the scalp, which can be altered by hair thickness)
   * Be dominant right-handed
   * Have a normal or corrected-to-normal vision
   * Be expected to comply with the protocol

Exclusion Criteria:

The project exclusion criteria are:

1. Conditions that may affect cortical oxygenation:

   * Be insomniac (insomnia severity index, ISI, higher than 15 based on rating at the medical screening) or night shift worker (based on anamnesis)
   * Be currently diagnosed with migraine (based on anamnesis)
   * Be currently diagnosed with hypo- or hyper-tension (based on evaluation of BP measure against medical norms at the medical screening)
   * Have an historical or current neural, cerebrovascular, cardiovascular, or respiratory disease (based on anamnesis)
   * Have a heavy usual consumption of caffeine-based beverages i.e., more than 5 servings of caffeinated coffee/colas or tea or 1 serving of caffeinated energy drinks per day
   * Be a regular smoker (regularly defined as greater than 2 cigarettes per week)
   * Participate in a vigorous physical activity requiring more than 6 metabolic equivalents e.g., hiking, jogging at 10 km/h or more, carrying of heavy loads, bicycling fast at 23 km/h or more, basketball, soccer, and tennis single, greater than 4 times 45 minutes per week
2. Conditions that may affect cognition or the mental fatigue

   * Take illicit drugs (for e.g., cannabis, heroin, and cocaine)
   * Have an average alcohol consumption greater than 2 standard drinks per day over a week for males, and greater than 1 standard drink per day over a week for females.

   One standard drink contains 10-12 g of ethanol. Examples of standard drinks are one beer can (300 ml), one glass of wine (100 ml) or one glass of schnaps (30 ml).
   * Have a psychiatric disorder or be currently diagnosed with anxiety or depression
   * Be pregnant (verified by a pregnancy test in urine dipstick format) or seeking to become pregnant or breast feeding
3. Have a hierarchal or family relationship with any of the research team members.
4. Currently participating in another interventional study.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will comprise of 36 healthy adults from 25 to 45 years old.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Modulation of cortical tissue oxygenation | Day 1
  Cortical tissue oxygenation parameters will be given by the concentration changes of oxygenated and deoxygenated hemoglobins measured with functional Near Infrared Spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Sélima Zahar, Master, Principal Investigator — Société des Produits Nestlé and Ecole Polytechnique Fédérale de Lausanne
Locations (1):
- Clinical Innovation Lab, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Access to the data will only be given to the academic laboratory hosting the aforementioned doctoral study. This concerns the Medical Image Processing laboratory, Ecole Polytechnique Fédérale de Lausanne.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will only be available from the preliminary to the last analysis performed (i.e. end of the study).
Access Criteria: A thesis agreement to cover the data protection has been agreed with the laboratory of the doctoral thesis director. The access to the data will be performed via secure directories of Société des Produits Nestlé.